CLINICAL TRIAL: NCT03814629
Title: Randomized Clinical Trial: Weifuchun Treatment on Precancerous Lesions of Gastric Cancer
Brief Title: Clinical Study of Weifuchun Treatment on Precancerous Lesions of Gastric Cancer
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: ShuGuang Hospital (Other)
Responsible Party: Principal Investigator, Mingyu Sun, Clinical Professor, ShuGuang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 42507214-9
Record Dates: First submitted 2018-08-30; First posted 2019-01-24 (Actual); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Chronic Atrophic Gastritis With Hyperplasia (Diagnosis)
Keywords: chronic atrophic gastritis; precancerous lesions of gastric cancer; Weifuchun; randomized clinical trial; mechanism
MeSH Terms: conditions — Disease; Gastritis, Atrophic | interventions — weifuchun; Vitamins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- precancerous lesions of gastric cancer (Other): 120 cases of chronic atrophic gastritis with intestinal metaplasia or dysplasia,It was randomly divided into 60 cases of treatment group and 60 cases of control group,treatment group was given Weifuchun tablets,The control group was given vitamin tablets.
  Interventions: Drug: Weifuchun

INTERVENTIONS:
Drug: Weifuchun — The treatment group（Weifuchun group）was given Weifuchun tablets, 4 tablets each time, 3 times a day, and 1 hour after meals. The control group(vitamin group) was given vitamin tablets (0.2 g), 4 tablets each time, 3 times a day, and 1 hour after a meal.
  Other Names: vitamin

SUMMARY:
Research purpose To elucidate the effect mechanism and clinical effective of weifuchun in the prevention and treatment of chronic atrophic gastritis and precancerous lesions of gastric cancer. From genes related to cell differentiation, proliferation, apoptosis, tumor invasion and metastasis, genes related to immune inflammation and immune escape and other possible aspects to elucidate the effective and mechanism of weifuchun's treatment on chronic atrophic gastritis, reversing precancerous lesions of gastric cancer.

DETAILED DESCRIPTION:
Clinical research abstract Title of Research Study：Randomized clinical trial: Weifuchun Treatment and mechanism on Precancerous Lesions of Gastric Cancer.

Main Responsibility Person: Mingyu Sun research center：Shuguang Hospital Affiliated to Shanghai University of Traditional Chinese Medicine Trial Objective：Observe the clinical efficacy and mechanism of Weifuchun in the treatment of chronic atrophic gastritis (CAG) and precancerous lesions of gastric cancer (PLGC) Therapeutic Schedule：Select 60 cases of chronic atrophic gastritis with intestinal metaplasia or dysplasia from and 60 cases of chronic atrophic gastritis without intestinal metaplasia or dysplasia at the Shuguang Hospital Affiliated to Shanghai University of Traditional Chinese Medicine. The treatment group was given Weifuchun tablets, 4 tablets each time, 3 times a day, and 1 hour after meals. The control group was given vitamin tablets (0.2 g), 4 tablets each time, 3 times a day, and 1 hour after a meal. The course of chronic atrophic gastritis with intestinal metaplasia or dysplasia group treatment is 24 weeks, the course of chronic atrophic gastritis without intestinal metaplasia or dysplasia is 12 weeks. The all patients'clinical symptoms, histopathology, gastroscopy, and physical and chemical examinations were compared between the two groups before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with chronic atrophic gastritis and precancerous lesions according to the pathological findings under gastroscope
2. Helicobacter pylori(-)

Exclusion Criteria:

1. Patients with Helicobacter pylori positive infection without radical treatment.
2. Patients with peptic ulcer, severe dysplasia or suspected malignant transformation.
3. Pregnant or lactating women and those who are pregnant and may not have effective contraception.
4. Patients with severe heart, lung, gallbladder, kidney, endocrine, hematopoietic system and neuropsychiatric diseases should not be included in this study.
5. Allergic constitution or known ingredients of this medicine.
6. Patients with other tumors.
7. Patients participating in other clinical trials within 1 month.
8. Patients with severe cirrhotic ascites and portal hypertension.
9. Other diseases that interfered with the study were deemed unsuitable for the patients included in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-08-01 (Actual); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
histopathology is assessing a change | the patients' were included into the clinical trials and after 24 weeks treatment.
  The all patients' histopathology will be evaluated two times, the first time is when the patients' are included into the clinical trials, the second time is after 24 weeks treatment in each group, patients' histopathology should be evaluated for comparison between two groups,at the same time patients' histopathology should be evaluated for comparison in each group.We use Total score of gastric mucosa pathology to assess the therapeutic effect,the patients' were included into the clinical trials and after 24 weeks treatment we through the Pathological classification of chronic atrophic gastritis work out Total score of gastric mucosa pathology.
  As follows:
  There are five pathology grade:Chronic inflammation,Active,Atrophy,intestinal metaplasia,dysplasia.
  Score 0 is normal;1 is mild; 2 is moderate;3 is severe;cumulative highest score is 15, cumulative lowest score is 0.The higher summed score, the more severe the pathological changes.
gastroscopy is assessing a change | the patients' were included into the clinical trials and after 24 weeks treatment.
  The all patients' gastroscopy gastric mucosa manifestations evaluation will be evaluated two times, the first time is when the patients' are included into the clinical trials, the second time is after 24 weeks treatment in each group, patients' gastroscopy gastric mucosa manifestations should be evaluated for comparison between two groups, at the same time patients' gastroscopy should be evaluated for comparison in each group.
  We use Gastric mucosa classification under gastroscope of chronic atrophic gastritis to assess the therapeutic effect,work out gastroscopy gastric mucosa manifestations integral.
  There are four Gastric mucosa classification under gastroscope of chronic atrophic gastritis: erythema,erosion,Intramucosal hemorrhage,bile regurgitation.Score 0 is normal;1 is mild; 2 is moderate;3 is severe;cumulative highest score is 12, cumulative lowest score is 0.The higher summed score, the more severe the pathological changes.
Clinical symptom score is assessing a change | the patients' were included into the clinical trials and after 24 weeks treatment.
  The all patients Clinical symptom assessment score when the patients' were included into the clinical trials and after 24 weeks treatment in each group. We use Clinical Symptom checklist to assess the therapeutic effect,work out Clinical Symptom integral. Clinical symptom mainly includes stomachache, acid reflux, burping, easy to hungry. Score 0 is frequency never;1 is occasionally; 2 is sometimes;3 is often; 4 is always. Summed highest score is 16, summed lowest score is 0.The higher summed score, the more severe the Clinical symptom.

SECONDARY OUTCOMES:
blood routine examination | the patients' were included into the clinical trials and after 24 weeks treatment
  The all patients ' blood routine examination(WBC,Hb,PLT) evaluation when the patients' were included into the clinical trials and after 24 weeks treatment in each group, this is for Clinical trial safety assessment.To assess the rate of abnormal blood routine examination(WBC,Hb,PLT) in each group.
liver function test | the patients' were included into the clinical trials and after 24 weeks treatment
  The all patients ' liver function test(ALT,Aspartate aminotransferase ,ALP) evaluation when the patients' were included into the clinical trials and after 24 weeks treatment in each group, this is for Clinical trial safety assessment.To assess the rate of abnormal liver function test(ALT,Aspartate aminotransferase ,ALP) in each group.
kidney function test | the patients' were included into the clinical trials and after 24 weeks treatment
  The all patients ' kidney function test(Cr,BUN) evaluation when the patients' were included into the clinical trials and after 24 weeks treatment in each group, this is for Clinical trial safety assessment.To assess the rate of abnormal kidney function test(Cr,BUN) in each group.

CONTACTS AND LOCATIONS:
Overall Officials: Mingyu Sun, doctor, Principal Investigator — Ethics Committee of Shuguang Hospital Affiliated to Shanghai University of Traditional Chinese Medicine

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bian Y, Chen X, Cao H, Xie D, Zhu M, Yuan N, Lu L, Lu B, Wu C, Bahaji Azami NL, Wang Z, Wang H, Zhang Y, Li K, Ye G, Sun M. A correlational study of Weifuchun and its clinical effect on intestinal flora in precancerous lesions of gastric cancer. Chin Med. 2021 Nov 20;16(1):120. doi: 10.1186/s13020-021-00529-9. PMID 34801051